CLINICAL TRIAL: NCT00309179
Title: A Single Arm Phase II Study of the Efficacy, Safety, and Biomarkers of Activity of E7820 Plus Cetuximab in Advanced Solid Tumors Preceded by a Run-In Study to Determine Safety of the Combination
Brief Title: A Phase II Study of the Safety and Efficacy of E7820 Plus Cetuximab in Colorectal Cancer, Preceded by a Run-in Study in Advanced Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7820-A001-204
Record Dates: First submitted 2006-03-29; First posted 2006-03-31 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Advanced Colorectal Cancer
Keywords: Advanced colorectal cancer
MeSH Terms: interventions — N-(3-cyano-4-methyl-1H-indol-7-yl)-3-cyanobenzene-sulfonamide; Cetuximab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: E7820 plus cetuximab

INTERVENTIONS:
Drug: E7820 plus cetuximab — Escalating doses from 40 mg/m^2 irinotecan plus E7820 in combination with cetuximab.

SUMMARY:
This study proposes to determine the safety of the administration of E7820 plus cetuximab and explore the MTD of the combination in a Phase Ib study. In addition, the efficacy of this combination will be explored in patients with colorectal cancer in the Phase II proof of concept phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* For Phase Ib, patients must have a histologically or cytologically confirmed malignant solid tumor for which no effective therapy is available or the patient must not be a candidate for standard therapy.
* For Phase II, patients must have a pathologically and histologically documented colorectal carcinoma that is inoperable and/or metastatic. These patients must also have at least one unidimensional measurable lesion according to the RECIST guidelines.
* Patients must have an ECOG Performance Status of 0-1.
* Patients must have a life expectancy of >= 3 months.
* Patients must be aged >= 18 years.
* Patients must have adequate renal function as evidenced by serum creatinine < 2 mg/dL and creatinine clearance > 40 mL/minute.
* Patients must have adequate bone marrow function as evidenced by ANC >= 1,500 /mm3 and platelets >= 100,000 /mm3.
* Patients must have adequate hepatic function as evidenced by liver function test abnormalities no greater than CTC grade 1 (bilirubin, alanine transaminase [ALT], and aspartate transaminase [AST]) unless increased LFTs are related to liver metastases in which case CTC grade 2 abnormalities acceptable.
* Patients must be willing and able to comply with the study protocol for the duration of the study.
* Patients must give written informed consent prior to any study-specific screening procedures with the understanding that the patient may withdraw consent at any time without prejudice.
* Patients may have received prior bevacizumab therapy as long as therapy has been discontinued for 4 weeks or longer.

Exclusion Criteria:

* Patients who have a history of previous Grade 2 or higher hypersensitivity to sulfonamide derivatives.
* Patients previously treated with cetuximab, or who have received prior treatment with any EGFR-related cancer therapy, either an approved or investigational agent.
* Patients with known sensitivity to murine monoclonal antibodies.
* Patients who have had radiation to >= 25% of their bone marrow (e.g., pelvic radiation) within 4 weeks prior to E7820 treatment.
* Patients who have not recovered from any clinically significant (Grade 3 or 4) chemotherapy, immunotherapy, or radiotherapy related toxicity at study entry (excluding neuropathy, infertility, or alopecia).
* Patients who have received investigational drugs or any other anti-neoplastic therapy within 28 days of E7820 treatment.
* Patients who have had major surgery within 4 weeks of study drug administration.
* Women who are pregnant or breast-feeding. Women of childbearing potential with either a positive pregnancy test at screening or no pregnancy test. Women of childbearing potential unless using adequate measures of contraception in the opinion of the Investigator (postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential).
* Fertile men and fertile women who are not willing to use contraception or fertile men or fertile women with a partner who is not willing to use contraception.
* Patients with brain or subdural metastases are not eligible except if they have completed local therapy and have discontinued the use of corticosteroids for this indication for at least one month before starting treatment with E7820. Any signs (eg, radiologic) and/or symptoms from their brain metastases must be stable for at least one month.
* Patients who have a positive history of human immunodeficiency virus, hepatitis B or active hepatitis C.
* Patients with severe uncontrolled intercurrent illness/infection (excluding malignancies).
* Patients with a history of unstable ischemic cardiac disease or more than Class II NYHA heart failure.
* Patients with a history of clinically significant arterial thrombosis or who have taken therapeutic doses of anticoagulants within the last 7 days.
* Patients who have pulmonary disease that puts them at risk of hemoptysis or bleeding diathesis. Head and neck cancer patients at risk for major vessel bleeding.
* Patients receiving therapeutics doses of anticoagulants.
* Patients with poorly controlled type I insulin-dependent diabetes or poorly-controlled type II insulin-dependent diabetes or a fasting blood glucose >10 mmol/L (200 mg/dL).
* Patients with significant comorbid disease or condition, which in the Investigator's opinion would exclude the patient from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-09-24 (Actual); Primary Completion 2009-12-14 (Actual); Study Completion 2017-02-13 (Actual)

PRIMARY OUTCOMES:
Objective tumor response (CR or PR) and disease control (CR, PR or SD) rates will be evaluated in this study based on RECIST criteria and modified WHO criteria. | The timing will be based on RECIST criteria and modified WHO criteria.

SECONDARY OUTCOMES:
Pharmacokinetics: Blood samples will be taken on Days 1, 2, and 15 during Cycle 1 and Day 1. Pharmacodynamics: Blood will be taken prior to dosing on Day 1, Days 1, 2, and 15 during Cycle 1 and Day 1. | Days 1, 2, and 15 during Cycle 1 and Day 1.

CONTACTS AND LOCATIONS:
Overall Officials: Eisai Medical Services, Study Director — Eisai Inc.
Locations (3):
- United States (2):
  - Los Angeles, California
  - Miami, Florida
- Edmonton, Alberta, Canada